CLINICAL TRIAL: NCT01634971
Title: Phase II Study of External Drainage Versus Internal Drainage of Pancreatic Duct With a Stent
Brief Title: External Drainage Versus Internal Drainage of Pancreatic Duct With a Stent After Pancreaticoduodenectomy (EDIDPD)
Acronym: EDIDPD
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CIH-WUQ-201205001; E2012010 (Other: E2012010)
Record Dates: First submitted 2012-07-03; First posted 2012-07-06 (Estimated); Last update posted 2016-02-17 (Estimated); Status verified 2013-01

CONDITIONS: Postoperative Fistula; Complications of Surgical and Medical Care: General Terms
Keywords: Postoperative pancreatic fistula(POPF);; Postpancreatectomy hemorrhage(PPH);; Delayed gastric emptying (DGE);; Bile leakage after pancreatic surgery;; Anastomotic leakage
MeSH Terms: conditions — Gastroparesis; Anastomotic Leak

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- External Drainage of pancreatic duct (No Intervention): External Drainage of pancreatic duct was used in PD.
- Internal Drainage of Pancreatic Duct (Experimental): the Intervention name is: Internal Drainage of Pancreatic Duct after pancreatomy, a stent was placed in the pancreatic duct, external drainage of the stent is defined as control group(the stent will be tans-abdomen and as a drainage of pancreatic fluid), and internal drainage of the stent is defined as interventional(or experimental) group, with the stent very short(2cm) and placed in jejunum.
  Interventions: Procedure: Internal Drainage of Pancreatic Duct after pancreatomy

INTERVENTIONS:
Procedure: Internal Drainage of Pancreatic Duct after pancreatomy — the Intervention name is: Internal Drainage of Pancreatic Duct after pancreatomy, a stent was placed in the pancreatic duct, external drainage of the stent is defined as control group(the stent will be tans-abdomen and as a drainage of pancreatic fluid), and internal drainage of the stent is defined as interventional(or experimental) group, with the stent very short(2cm) and placed in jejunum.
  Arms: Internal Drainage of Pancreatic Duct

SUMMARY:
Postoperative pancreatic fistula (POPF) and other surgical complications are common after pancreatoduodenectomy (PD) and POPF is a major complication. The drainage of pancreatic duct is important and a stent is usually placed in the operation, but it is still controversial whether the stent drainage is internal or external.

DETAILED DESCRIPTION:
The current study is to compare the rate of Postoperative pancreatic fistula(POPF) and other surgical complications after pancreatoduodenectomy (PD).

ELIGIBILITY:
Inclusion Criteria:

* Age more than 18 years.
* Received pancreatoduodenectomy.
* Informed consent has been signed.

Exclusion Criteria:

* Age less than 18 years
* Emergency surgery
* Past history of pancreatic surgery.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2012-05; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
the rate of Postoperative pancreatic fistula within 2 weeks after operation | within 2 weeks after operation
  Postoperative pancreatic fistula (POPF) is defined as a drain output of any measurable volume of fluid on or after postoperative day 3 with an amylase content greater than 3 times the serum amylase activity.

SECONDARY OUTCOMES:
the rate of postoperative Surgical Complications | 2 weeks after operation
  the rate of Postpancreatectomy hemorrhage(PPH);Delayed gastric emptying (DGE); Bile leakage after pancreatic surgery;Anastomotic leakage

CONTACTS AND LOCATIONS:
Overall Officials: Qiang WU, MD. Ph.D., Study Chair — Tianjin Medical University Cancer Institute and Hospital
Locations (1):
- Tianjin Medical University Cancer Institute and Hospital, Tianjin, Tianjin Municipality, China